CLINICAL TRIAL: NCT03270319
Title: Evaluation of Three Dimensional Echocardiography in Critical Care Medicine
Acronym: 3DICU
Status: Terminated | Type: Observational
Why Stopped: Study team members moved away
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 16032016
Record Dates: First submitted 2016-03-17; First posted 2017-09-01 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Shock
Keywords: Measurement of cardiac output
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patient: Critically ill patients in our adult intensive care unit with the following characteristics:
  * advanced hemodynamic monitoring in place including pulmonary artery catheter and arterial catheter
  * intubated or tracheostomy in place
  * echocardiography requested by the treating physician
  * intervention of interest: hemodynamic assessment done by echocardiography and thermodilution (pulmonary artery catheter)

SUMMARY:
Comparison of volumetric measurements obtained by three dimensional echocardiography with measurements obtained by thermodilution using a pulmonary artery catheter in the intensive care unit.

DETAILED DESCRIPTION:
Prospective, observational study evaluating three dimensional echocardiography for measuring hemodynamic variables versus the current gold standard (pulmonary artery catheter).

Critically ill patients with a severly compromised circulation due to a shock state with an advanced hemodynamic monitoring in place and the need for echocardiographic evaluation will be included.

While performing an echocardiography study stroke volume measurements using the bolus method for thermodilution will concomittantly be measured.

In case of insufficient image quality we are planning to use SonoVue echo contrast. Once the image quality has improved we will repeat the stroke volume measurements with the bolus thermodilution method while performing the echocardiography.

The acquired echocardiography loops will then be analysed and measured offline once deferred consent has been obtained. We will then compare the echocardiographic measurements with the measurement obtained by the pulmonary artery catheter (bolus method) - since this is the current reference method.

ELIGIBILITY:
Inclusion Criteria:

* advanced hemodynamic monitoring with pulmonary artery catheter and arterial catheter in place
* patient intubated or tracheostomy in place
* clinical indication for performing an echocardiography
* ongoing sedation requirement

Exclusion Criteria:

* Heart rhythm other than sinus rhythm or paced atrial rhythm
* Known allergy to sulphur-hexafluoride (SonoVue©)
* Artificial heart valves in place
* Any form of mechanical cardiac assist
* contraindication to performing a transesophageal echocardiography
* presence of significant cardiac valve regurgitation
* presence of an intracardiac shunt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult intensive care patients treated in our intensive care unit with current hemodynamic unstable condition.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Comparison of stroke volume measurement with three dimensional echocardiography to stroke volume measurement by thermodilution | through study completion, an average of 1 year
  The stroke volume of three to six heart beats will be measured after having performed an echocardiographic study. The stroke volume by thermodilution will be measured during the individual examination.

SECONDARY OUTCOMES:
Feasibility of right ventricular pressure volume loops | through study completion, an average of 1 year
  Off-line analysis of pressure time curve for right ventricle using data from pulmonary artery catheter and volume time curve from echocardiographic data. Assessment of feasibility to combine these two curves to a pressure volume loop.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bloch, MD, Principal Investigator — Department of intensive care medicine, Luzerner Kantonsspital
Locations (1):
- Department for Intensive Care Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No